CLINICAL TRIAL: NCT00231101
Title: Quetiapine Decreases Smoking in Patients With Chronic Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arthur P. Noyes Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: NSH Protocol 03-08
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2005-09

CONDITIONS: Smoking Behavior in Schizophrenia
Keywords: Smoking; Schizophrenia
MeSH Terms: conditions — Smoking; Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine

SUMMARY:
A single-blind switching study in which forty subjects currently being treated with risperidone will be randomly assigned to either stay on risperidone or switched to quetiapine. Various behavioral and biological measures will be used to compare smoking behavior over time in these two groups.

DETAILED DESCRIPTION:
STUDY SYNOPSIS

Study Design

Number of subjects enrolled: Forty patients (Two groups - 20 each)

Number of centers: One

Study design: Single-blind, Switching Paradigm

Extension: None specifically, although patients who do have a good clinical response to the treatment will probably be maintained on their medication at the discretion of their treating psychiatrist through normal hospital channels and, therefore, if desired, it would be possible to formally re-evaluate their condition at some later time.

Duration of study:

Total duration of subject participation: 14 weeks Duration of each study phase: Screening: 1-7 days Lead-in treatment with risperidone: 2 weeks Switching phase: 50% of the patients will be switched over a two-week period to quetiapine Active two group treatment: 12 weeks

Visit interval or frequency: variable, depending on measurement Weekly - dispensing drug & treatment team meeting Bi-weekly - labs & certain side effect ratings Monthly - efficacy measures and side effect ratings Baseline, Week 6 & Week 12 - cognitive measures

Recruitment/enrollment duration: Approximately 18 months

Subject Population

Specific subject population/disease state/disorder being studied:

Patients with DSM-IV schizophrenia (all sub-types, including schizoaffective disorder) who are active heavy smokers (at least one pack of cigarettes per day) will be recruited. To be included each patient will need to have received an adequate dose and duration of risperidone treatment (monotherapy of at least 6 mg total daily for three months or more) and who had a less-than-optimal response treatment. Specifically, a less-than-optimal response to risperidone is defined as a Total PANSS Score of 60 or more. Additionally, we will not enroll clinically stable patients who are satisfied with their ongoing treatment or patients judged to be treatment refractory (using Kane's criteria).

Subject setting: both Norristown State Hospital inpatients and those enrolled in a partial hospital program will be recruited.

Partial: On the grounds of Norristown State Hospital are three partial hospital programs administered by the Montgomery County Office of Mental Health. These are highly structured programs that will allow us to recruit subjects who are outpatients but living in well-supervised programs.

Inpatient: Norristown State Hospital 1001 Sterigere Street Norristown, PA 19401

Study drug and dosing:

Flexible: To be enrolled, all patients will have had an adequate treatment of risperidone (defined as monotherapy of at least 6 mg total daily for three months or more) prior to enrollment. For those switched from risperidone to quetiapine, it is expected this cross-titration will take two weeks (longer titration may be used if necessary due to higher levels of risperidone). By the end of the first week, the risperidone will be reduced by 50% of the patient's original dosage, with the target dose of quetiapine being 400 mg total daily dose at the end of the first week. By the end of the second week of titration, the risperidone will be discontinued, and the treating psychiatrist will continue to increase the quetiapine to the target of 600 mg total daily dose based on his/her clinical judgement, then to reach 800 mg total daily dose by the end of the fourth week. A lower dose will be possible due to emergent side effects, but any patient not able to tolerate at least 400 mg/day of quetiapine will be dropped from the study. Quetiapine will be dosed BID.

Comparator(s) and dosing:

Flexible: As stated above, all patients will have had an adequate treatment of risperidone prior to enrollment. It is expected that the majority of those patients remaining on risperidone will continue to be treated at the 6 mg/day dose, although their treating psychiatrist will be able to suggest a lower dose due to side effects or increase the dose as necessary for greater efficacy. Any patient requiring less that 4 mg/day or more than 10 mg/day will be dropped from the study. While risperidone is usually dosed on a once per day basis, throughout the switching phase of the study it will be dosed BID. The possibility exists that once/daily versus twice/daily dosing could be a factor that influences medication compliance rates between the groups, and a source of bias. Twice/daily dosing for both groups would also help to insure the blinding of the raters.

It is important to note that no formal consensus exists regarding the milligram-to-milligram equivalency of risperidone and quetiapine. However, based on personal communication with Herbert Meltzer, M.D., it seems that these dose ranges are thought to be comparable (1 mg risperidone = approximately 100 mg quetiapine). Thus, the ideal comparison of 6 mg/day risperidone to 600 mg/day quetiapine should avoid criticism, although, the final group mean doses will finally be determined on the basis of individual patient treatment response and emergent side effects.

Other treatments or programs:

There will be no other study related treatment programs, although each patient (whether inpatient or partial hospital patient) will continue to receive their usual hospital or clinic care on a regular basis. It is critical to note, however, that any patient receiving ancillary behavioural, psycho-educational, or pharmacologic treatment for smoking cessation will not be enrolled due the inherent bias and/or uncontrolled variance introduced by additional treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male or female) between 18-65 years of age must be diagnosed as having DSM-IV schizophrenia (any subtype including schizoaffective disorder).
2. Patients must have shown a less-than-optimal clinical response to an adequate course of risperidone treatment and must be willing to agree to the possibility of receiving quetiapine as an alternative treatment for their mild to moderate psychotic symptoms. We define an adequate course of treatment as three or more months of at least 6 mg/day of risperidone. We define less-than-adequate treatment as a Total PANSS Score of 60 or more.
3. Patients must be active cigarette smokers. We define active cigarette smoking as patients who consume one pack of cigarettes or more per day. Although there is no standard for defining active cigarette smokers, it has been our experience that the high rate of smoking activity on the hospital wards can have the effect of small elevations in cotinine levels even among "non-smoking" patients through second hand smoke. Therefore, we want to insure that we enroll "heavy" smokers.
4. Patients must be able to fully participate in the informed consent and HIPAA process, or have a legal guardian able to participate

Exclusion Criteria:

1. Patients who have had an adequate clinical response to risperidone and are considered by themselves or their treating psychiatrist to be clinically stable.
2. Patients who are judged to be treatment refractory, which we define as documented treatment failure with 3 FDA-approved antipsychotic medications administered for an adequate duration in a sufficient dosage (6 or more weeks of 1000 mg/day chlorpromazine equivalents).
3. Patients at the time of screening who have clinically significant akathisia (Barnes global score >2), Parkinsonian symptoms symptoms (Simpson Angus total score >3), or significant EPS (indicated by treatment with benztropine, lorazepam or propranolol).
4. ECG abnormalities consistent with significant or acute cardiac disease.
5. History of significant or unstable hypertension during the screening examination outside the range from 90/60 to 140/90, or a pulse outside of the range of 60 to 100 beats per minute.
6. Any history of seizures or primary CNS disease (other than tardive dyskinesia or extrapyramidal symptoms from psychotropic medications), comatose states, bone marrow depression, significant cardiovascular, renal or hepatic disease, brain trauma, chronic obstructive lung disease and/or pulmonary emphysema, or a mental deficiency.
7. Active drug or alcohol addiction within the past 3-month period.
8. Symptoms of significant physical illness in the 4-week period prior to enrollment, excluding mild upper respiratory or gastrointestinal disorders.
9. Clinical laboratory findings that indicate the presence of a pathological condition in the judgment of the principal investigator.
10. Having received any investigational drug in the 4 weeks preceding the study.
11. Pregnant or lactating patients are excluded. Pregnancy must be excluded by laboratory tests prior to beginning the study. Female patients judged to have potential for pregnancy (sexually-active females who do not use an approved form of contraception) will be excluded.
12. At serious suicidal risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2006-06

PRIMARY OUTCOMES:
The Fagerstrom Test for Nicotine Dependence,weekly measures of expired CO and blood levels of cotinine. The endpoints for assessing nicotine receptor activation will include: the auditory P50, visuospatial working memory, and the CPT.
Changes in psychopathology will be performed monthly PANSS, CGI, and the SANS.
EPS will be measured weekly using the NRS, and the Barnes Akathisia Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Josiassen, Ph.D., Principal Investigator — Arthur P. Noyes Research Foundation
Locations (1):
- Arthur P. Noyes Research Foundation, Norristown, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.noyesfoundation.net